CLINICAL TRIAL: NCT00870493
Title: The Safety and Short-Term Efficacy of Aliskiren in the Treatment of Immunoglobulin A Nephropathy - A Randomized Cross-Over Study
Brief Title: Aliskiren for Immunoglobulin A (IgA) Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AIgA
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: IgA Nephropathy
Keywords: proteinuria; renal failure; glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria; Renal Insufficiency; Glomerulonephritis | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): each subject will receive oral aliskiren 300 mg/day for 16 weeks, followed by a washout period of 4 weeks, then crossed over to placebo for another 16 weeks
  Interventions: Drug: Aliskiren; Drug: Placebo
- II (Active Comparator): each subject will receive placebo for 16 weeks, followed by a washout period of 4 weeks, then crossed over to oral aliskiren 300 mg/day for another 16 weeks
  Interventions: Drug: Aliskiren; Drug: Placebo

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 300 mg daily oral
Drug: Placebo — starch tablet, 300 mg/day

SUMMARY:
Immunoglobulin A (IgA) nephropathy is the most common type of primary glomerulonephritis in the world. Current treatment with angiotensin converting enzyme (ACE) inhibitor and angiotensin receptor blocker (ARB) is not entirely effective. Aliskiren, a direct renin inhibitor, acts on the rate limiting step of the renin-angiotensin axis. In addition to lowering the blood pressure, recent study in diabetic nephropathy suggests an independent anti-proteinuric effect. The investigators plan to conduct a randomized placebo-control cross-over study to evaluate the safety and efficacy of aliskiren in the treatment of IgA nephropathy. The investigators plan to recruit 57 patients with biopsy-proven IgA nephropathy and persistent proteinuria despite conventional therapy. They will be randomized to aliskiren for 16 weeks or no treatment, followed by cross over to the other arm after a washout period. Proteinuria, albuminuria, renal function, serum and urinary markers will be quantified. This study will explore the potential anti-proteinuric effect of aliskiren in the treatment of IgA nephropathy, which has no specific treatment at present.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* requires anti-hypertensive therapy
* renal biopsy within the past 3 years and confirmed the diagnosis of IgA nephropathy
* proteinuria > 1 g/day (or proteinuria > 1 g/g-Cr) in 3 consecutive samples within 12 weeks despite ACE inhibitor or ARB treatment for at least 3 months
* estimated glomerular filtration rate > 30 ml/min/1.73m2
* willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* Patients who are diabetic, and patients with systemic diseases that may cause IgA nephropathy or another nephropathy.
* Pregnancy, lactating or childbearing potential without effective method of birth control
* Severe gastrointestinal disorders that interfere with their ability to receive or absorb oral medication
* History of malignancy, including leukemia and lymphoma within the past 2 years
* Systemic infection requiring therapy at study entry
* Any other severe coexisting disease such as, but not limited to, chronic liver disease, myocardial infarction, cerebrovascular accident, malignant hypertension
* History of drug or alcohol abuse within past 2 years
* Participation in any previous trial on aliskiren or other renin inhibitor
* Previous treatment with fish oil, steroid, cytotoxic agents, or aldosterone antagonist
* History of treatment with other drugs that may affect proteinuria within past 2 years
* Patients receiving treatment of corticosteroid
* On other investigational drugs within last 30 days
* History of a psychological illness or condition such as to interfere with the patient's ability to understand the requirement of the study
* History of non-compliance
* Known history of sensitivity or allergy to aliskiren or other renin inhibitor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
change in the degree of proteinuria | 16 weeks

SECONDARY OUTCOMES:
rate of decline of estimated GFR | 16 weeks
change in serum and urinary inflammatory markers | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Szeto CC, Kwan BC, Chow KM, Leung CB, Li PK. The safety and short-term efficacy of aliskiren in the treatment of immunoglobulin a nephropathy--a randomized cross-over study. PLoS One. 2013 May 10;8(5):e62736. doi: 10.1371/journal.pone.0062736. Print 2013. PMID 23675422